CLINICAL TRIAL: NCT06385067
Title: Prospective, International Multicenter Clinical Study Evaluating the Safety and Efficacy of the Biolimus Coated Coronary Artery Balloon Dilation Catheter (BioAscend) in the Treatment of Primary Coronary Artery Disease in the Real World
Brief Title: Treatment of Primary Coronary Artery Vascular Lesions With Biolimus Coated Coronary Balloon Dilation Catheter
Status: Not yet recruiting | Type: Observational
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: JW-PM-DCB-2024
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Use at least one Biolimus coated coronary balloon dilation catheter (BioAscend) to treat primary in situ coronary artery vascular disease with a diameter of 2.0 mm-2.75 mm regardless of the number of blood vessels, the length and number of treated lesions.
  Interventions: Device: Biolimus Coated Coronary Artery Balloon Dilation Catheter

INTERVENTIONS:
Device: Biolimus Coated Coronary Artery Balloon Dilation Catheter — Patients with Coronary Artery Disease will be treated with Biolimus Coated Coronary Artery Balloon Dilation Catheter

SUMMARY:
The purpose of the study was to further evaluate the long-term safety and efficacy of the Biolimus Coated Coronary Artery Balloon Dilation Catheter in the real world.

The study population was patients with primary coronary vascular lesions with a blood vessel diameter of 2.0mm-2.75mm.

DETAILED DESCRIPTION:
Study Design:

1. Prospective, international multi-center clinical study;
2. It is planned to recruit 300 subjects in China and a total of 100 subjects in Indonesia and Thailand who meet the criteria for study inclusion to use at least one Biolimus coated coronary balloon dilation catheter (BioAscend) to treat primary in situ coronary artery vascular disease with a diameter of 2.0mm-2.75mm regardless of the number of blood vessels, the length and number of treated lesions;
3. In the study, subgroups of long lesions, bifurcation lesions, and acute myocardial infarction were set up, and subjects who met the definition were directly entered into the subgroup analysis.
4. Register and collect data using the EDC system;
5. Enrollment method: competitive enrollment;
6. Follow-up time points: postoperative to before discharge, 30 days, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Primary coronary artery stenosis with a vessel diameter of 2.0 mm to 2.75 mm;
* Patients with residual stenosis of ≤ 30 percent after pretreatment and ≤ type B dissection; Patients who voluntarily participate in and sign the informed consent form, and who are willing to undergo follow-up as required by the protocol.

Exclusion Criteria:

* Pregnant or lactating females;
* Patients with cardiogenic shock;
* Patients with severe congestive heart failure or severe heart failure with NYHA class IV;
* Patients with severe valvular heart disease;
* Patients with a life expectancy of less than 24 months or factors that make clinical follow-up difficult;
* Patients who are considered unsuitable for inclusion by the investigator for other reasons.
* Those who are known to be allergic to melcrolimus and contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruit 300 subjects in China and a total of 100 subjects in Indonesia and Thailand who meet the criteria for study inclusion to use at least one Biolimus coated coronary balloon dilation catheter (BioAscend) to treat primary in situ coronary artery vascular disease with a diameter of 2.0mm-2.75mm regardless of the number of blood vessels, the length and number of treated lesions;
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure rate (TLF) | 12 months after surgery
  Target lesion failure rate (TLF) at 12 months after surgery, including cardiogenic death, target vascular myocardial infarction, and clinically symptom-driven target lesion revascularization (CD-TLR)

SECONDARY OUTCOMES:
Interventional success rate | Immediately after operation
  Including device success rate, pathogenic power and clinical success rate
Device-related cardiovascular clinical composite endpoint | From postoperative to before discharge, day 30, month 6, month 12, month 24
  Device-related cardiovascular clinical composite endpoints from postoperative to pre-discharge, day 30, month 6, month 12, and month 24, including cardiac death, target vessel myocardial infarction, and clinically symptom-driven target lesion revascularization (excluding elective interventional therapy)Device-related cardiovascular clinical composite endpoints from postoperative to pre-discharge, day 30, month 6, month 12, and month 24, including cardiac death, target vessel myocardial infarction, and clinically symptom-driven target lesion revascularization (excluding elective interventional therapy)
Patient-related cardiovascular clinical composite endpoint | From postoperative to before discharge, day 30, month 6, month 12, month 24
  Patient-related cardiovascular clinical composite endpoints including all-cause mortality, all myocardial infarction, and any revascularization (excluding elective interventional therapy) from postoperative to pre-discharge, day 30, month 6, month 12, and month 24
Major adverse cardiac events (MACEs) | From postoperative to before discharge, day 30, month 6, month 12, month 24
  Including cardiac death, myocardial infarction, and target lesion revascularization (TLR) at postoperative to pre-discharge, day 30, month 6, month 12, and month 24.
Incidence of thrombotic events as defined by ARC | From postoperative to before discharge, day 30, month 6, month 12, month 24
  Including identified, probable, and unexcluded thrombosis in the acute, subacute, and late periods acute, subacute, and late Defined, probable, and non-excluded thrombosis within the segment

CONTACTS AND LOCATIONS:
Overall Officials: Lang Li, Principal Investigator — First Affiliated Hospital of Guangxi Medical University

IPD SHARING:
Plan to Share IPD: No